CLINICAL TRIAL: NCT04057404
Title: Smartphone Twelve Lead Electrocardiogram Utility In ST Elevation Myocardial Infarction
Acronym: ST LEUIS
Status: Completed | Type: Observational
Sponsor: INTEGRIS Baptist Medical Center (Other)
Responsible Party: Principal Investigator, Charles Bethea, Principal Investigator, INTEGRIS Baptist Medical Center
Other Study IDs: INT15-017
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: ST Elevated Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Alivecor Heart Monitor
  Other Names: Smartphone ECG

SUMMARY:
The primary objective is to determine if the Smartphone electrocardiogram (ECG) is an acceptable replacement for a standard ECG in the identification of ST elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
Toward this objective, this study involves the following:

* Obtain simultaneous recordings of a standard 12-lead ECG and the iPhone "12-lead equivalent" ECG on patients presenting with chest pain in which the STEMI protocol was activated.
* Obtain simultaneous recordings of a standard 12-lead ECG and the iPhone "12-lead equivalent" ECG on patients presenting to the Emergency Department for evaluation of chest pain, not necessarily presenting with STEMI.
* Reading of ECGs (standard 12-lead and iPhone) by three independent cardiologists, who are blinded to the initial clinical ECG readings, the type of ECG equipment used, and the patient's clinical information.
* Assess the operational feasibility of using the Smartphone to obtain "12-lead equivalent" ECG recordings in patients suspected to have STEMI, and
* Determine the possibility of pooling the data obtained from this study with data from other institutions conducting identical studies, and developing a future IRB-approved protocol and statistical analysis plan to compare the sensitivity, specificity, positive predictive value and the negative predictive power of the iPhone ECG, using a paired standard 12-lead ECG as the gold standard.

There will be no therapeutic interventions. A single research-related procedure will be required, i.e. an iPhone ECG. Effort will be made to ensure that the performance of this procedure will not delay any treatment and/or diagnostic procedures that are part of usual or specialized care that the patient requires. Effort will be made to enroll 1 STEMI patient for every 2 non-STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age.
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures (patient or legally acceptable representative).
* Symptoms of chest pain upon presentation at the INTEGRIS Baptist Medical Center Emergency Department

Exclusion Criteria:

* Inability or refusal of the patient and/or the patient's legally-acceptable representative to provide written informed consent for any reason.
* Other conditions that in the opinion of the Principal Investigator or Co-Investigator(s) may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients, >18 years old, who are seen for chest pain, and/or patients for whom the STEMI protocol has been activated, will be screened for this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Determine the number of agreements in diagnoses (STEMI vs. non-STEMI) between the standard 12-lead ECG and the iPhone "12-lead equivalent" ECG | 10 Weeks
  Number of Agreements

CONTACTS AND LOCATIONS:
Locations (1):
- INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No